CLINICAL TRIAL: NCT05251025
Title: Comparative Effects of Myofascial Release and Sustained Stretching on Hamstring Flexibility in Spastic Cerebral Palsy Children
Brief Title: Myofascial Release and Sustained Stretching in Spastic CP Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0220 Iqra Khalid
Record Dates: First submitted 2022-02-20; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy
Keywords: Spastic cerebral palsy; Passive Sustained Stretching; Myofascial Release; MAS; Goniometer
MeSH Terms: conditions — Cerebral Palsy | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive sustained stretching (Experimental): Passive sustained stretching along with conventional treatments
  Interventions: Other: Passive sustained stretching
- Myofascial Release (Experimental): Myofascial Release Technique along with conventional treatments
  Interventions: Other: Myofascial Release

INTERVENTIONS:
Other: Passive sustained stretching — The Group A received Passive Stretching Technique. Along with the Passive Stretching Technique, this group also received certain conventional treatments which included resistive exercises, gait training exercises, bridging and exercises in other functional positions were also undertaken by the included individuals.
  All the exercises mentioned above were performed for 30 minutes and there was not any specific division of time for all these mentioned activities. The patients used to perform these conventional treatments and exercises on their motor control basis. The exercises were performed for 30 minutes and been done for 5 days in a week for consecutive 6 weeks.
  Arms: Passive sustained stretching
Other: Myofascial Release — The Group B received Myofascial Release Technique and along with conventional treatments. The Myofascial Release Technique for hamstrings was given to the patient in prone position. The technique was applied either by the crossed hands or thumbs. This total treatment was given for 30 minutes consecutively. After the technique the Myofascial structures were stretched and then were hold for straight 120 seconds so that the tissues get softened. The technique was given to patients with 6 repetitions and with a hold for 120 seconds. The treatment was continued for 5 days a week for straight 6 weeks.
  Arms: Myofascial Release

SUMMARY:
The aim of this research was to find and compare the effects of Myofascial Release Technique and Passive Sustained Stretching on Hamstrings Flexibility in Children with Spastic Cerebral Palsy.

DETAILED DESCRIPTION:
Randomized Clinical Trials done at DHQ Sahiwal. 26 spastic CP children of age 6-12 years were taken by random sampling technique from DHQ Sahiwal. 13 were allocated to each group. Study duration was of 6 months. Sampling technique applied was non probability convenience sampling technique Group A received Passive Sustained Stretching along with conventional treatment. Whereas Group B received MFR along with conventional treatment. Both these groups received treatment for 6 weeks. The baseline and post treatment score of MAS, Goniometer (AKET to measure popliteal angle) and GMFCS -88 were evaluated. Data analysis was done by using the SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 6 to 12 years were included.
* Both genders were included.
* Ambulatory subjects with or without ambulatory aids.
* Diagnosed children with Spastic CP.
* CP patients with grade 3 on modified Ashworth scale for hamstrings were included

Exclusion Criteria:

* Children with visual or auditory defects.
* Children with cognitive dysfunction.
* Subjects who had severe limitations in passive range of motion at lower extremities specially hamstrings due to surgery or any other complication.
* Children with other types of Cerebral Palsy such as Ataxic CP, Dyskinetic CP etc.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | 6th week
  Modified Ashworth scale is one of the most internationally accepted clinical tool that is to measure the increased tone in the muscles. Ashworth Scale in 1964 was published by Bryan Ashworth. This clinical tool has been used as a method for grading spasticity, especially in patients with Cerebral Palsy, Multiple sclerosis etc. The reliability of Modified Ashworth Scale is(ICC+=0.686).
Gross Motor Function Classification System | 6th week
  The Gross Motor Function Classification System (GMFCS-88) is a five-level system that is basically is considered as a standardized method to explain gross motor function in CP Children. This GMFCS is used in CP Children with age ranging from 1 to 12 years. The basic focus in this tool is the sitting and walking of the CP Children. This classification system can simply be merged into medical practice. This will help to make assessments of the affected children. It also shows major or clear differences in the gross motor functions of Cp children that are impactful in the daily activities. the intra-rater and inter-rater reliability of GMFCS is 0.98 and 0.97 respectively
Active Knee Extension Test | 6th week
  For Active Knee Extension Test that helped to measure popliteal angle the patient was asked to lie supine on the examination table with hip and the knee flexed to 90 degrees and the test was done on both legs alternatively. The examiner then supported the testing thigh so that it remained vertical and asked the patient to extend the knee actively while the contralateral leg remained extended. This active knee extension was done voluntarily. After this, the examiner held that knee extension for 5 seconds to support and keep the stretch to find the point of maximum resistance to ensure the exact readings. To measure the readings, the examiner placed a 360 degrees goniometer on the landmarks being marked for taking the readings. The landmarks used as reference for goniometer were greater trochanter of the femur and lateral malleolus of the tibia.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, PPDPT, Principal Investigator — Riphah International University
Locations (1):
- District Head Quarter Hospital, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No